CLINICAL TRIAL: NCT00655434
Title: HerpeSelect® Express Rapid Test Study Protocol Sexually Active Adult Population
Brief Title: HerpeSelect® Express Rapid Test Study Protocol: Sexually Active Adult Population
Status: Completed | Type: Observational
Sponsor: Focus Diagnostics, Inc. (Industry)
Responsible Party: John Hurrell/Vice President General Manager, Focus Diagnostics, Inc.
Other Study IDs: 06-001-RT0920G Rev:03/07/08
Record Dates: First submitted 2008-04-02; First posted 2008-04-09 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Herpes Simplex Virus 2
Keywords: Herpes simplex virus 2; HSV 2; Antibody status to Herpesvirus 2, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SAA: Sexually Active Adults- Intercourse in the last twelve months with at least one sexual partner. Subjects must be ≥ 18 years old. No more than 60% of one gender.

SUMMARY:
This study is designed to compare the performance of the Focus Diagnostics' HerpeSelect® Express, a Herpes Simplex Virus 2 Rapid Test, to a currently marketed device. The intent is to show the rapid test device is comparable to the currently marketed device. HerpeSelect® Express is a rapid test intended for qualitatively detecting the presence or absence of human IgG class antibodies to herpes simplex virus type 2 (HSV-2) in human whole blood (capillary).

DETAILED DESCRIPTION:
The objective of this study is to establish the performance characteristics of the Focus Diagnostics (Focus) HerpeSelect® Express based on comparison to the Focus Diagnostics' HerpeSelect® 2 ELISA IgG (K021486). The Focus HerpeSelect® 2 ELISA IgG device is intended for qualitatively detecting the presence or absence of human IgG class antibodies to HSV-2 in human sera. Positive samples in either the HerpeSelect® 2 ELISA IgG or HerpeSelect® Express will be tested in the HerpeSelect® Immunoblot (K000238).

This external study along with in-house analytical studies will demonstrate the efficacy of the HerpeSelect® Express Rapid Test device as an aid in screening for pregnant women or sexually active adults as in the presumptive diagnosis of HSV-2 infection for point-of-care testing sites as well as hospital/clinics and reference laboratories. Independent sites in the Southeastern, Western, Eastern, and Pacific Northwestern U.S. will test subjects with the HerpeSelect® Express Rapid Test. Sera from those patients will be tested at Focus Diagnostics Reference Laboratory in the HerpeSelect® 2 ELISA IgG. Discrepants between HerpeSelect® Express Rapid Test and HerpeSelect® 2 ELISA IgG may be tested in the HerpeSelect® Immunoblot IgG assay.

Test subjects will be from three patient populations: 375 sexually active adults, 375 pregnant women, and 100 low prevalence adults. Two samples types will be collected from each subject: capillary whole blood and serum. These samples types will be tested with both the HerpeSelect® Express Rapid Test and HerpeSelect® 2 ELISA IgG.

ELIGIBILITY:
Inclusion Criteria:

* Sexually Active Adults - Intercourse in the last twelve months with at least one sexual partner.
* Subjects must be ≥ 18 years old.
* No more than 60% of one gender.

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community based research clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Compare serological status to predicate device | End of study

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Clinical Research, Burbank, California, United States